CLINICAL TRIAL: NCT07349901
Title: Predicting Hospital Readmission for Surgical Patients Using Deep Learning Models With Smart Watch and Smart Ring Sensors Data
Status: Not yet recruiting | Type: Observational
Sponsor: Getúlio Vargas University Hospital (Other Government)
Collaborators: Universidade Federal do Amazonas (Other); Samsung Eletrônica da Amazônia Ltda (Unknown)
Responsible Party: Sponsor
Other Study IDs: 91090825.8.0000.5020; Convênio No 03/2025 (Other Grant/Funding Number: SAMSUNG ELETRÔNICA DA AMAZONIA)
Record Dates: First submitted 2025-12-02; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Patient Readmission
Keywords: Hospital Readmission; Postoperative Complications; Artificial Intelligence; Machine Learning; Wearable Electronic Devices; Physiological Monitoring; Sleep Disorders; Surgical Procedures, Operative; Perioperative Care; Amazon Region; Predictive Modeling
MeSH Terms: conditions — Postoperative Complications; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hospital readmissions are an important measure of healthcare quality and safety. These events create a substantial burden for patients, families, and health systems because they may increase costs, extend recovery time, and lead to more serious postoperative complications. Predicting which patients are at higher risk of readmission remains difficult, as many complications begin silently and are not easily identified in routine clinical evaluations.

This study aims to evaluate whether artificial intelligence (AI) can help predict hospital readmissions in surgical patients by analyzing physiological and behavioral data collected before and after surgery. To achieve this, participants will use wearable devices-specifically a smartwatch and a smart ring-capable of continuously monitoring health biomarkers such as heart rate, electrocardiogram (ECG), oxygen saturation, sleep patterns, blood pressure trends, body composition through bioimpedance, and stress indicators. These devices are provided through a technology partnership and sponsorship from Samsung, which supports the study with advanced health technologies.

This is a prospective, single-center cohort study conducted at the main tertiary hospital in the state of Amazonas. Approximately 225 to 300 adults undergoing medium- or large-scale elective surgeries will be invited to participate over a 25-month period. All participants will provide informed consent. After enrollment, the study will collect demographic information, preoperative assessments, validated sleep questionnaires, comorbidity indexes such as the Charlson Comorbidity Index, laboratory exams, pulmonary function tests, intraoperative and postoperative data, and hospital discharge information.

Participants will be continuously monitored using wearable devices during their hospital stay-including the first 48 hours in the intensive care unit when applicable-and for 30 days after hospital discharge. These physiological data will be integrated with clinical and laboratory information to create a comprehensive dataset.

The primary objective is to develop and test artificial intelligence models capable of predicting 30-day hospital readmission following elective surgery. Both deep learning approaches and classical machine-learning techniques will be evaluated. By analyzing large volumes of continuous physiologic data, these models may identify early signs of postoperative deterioration that would otherwise go unnoticed.

If successful, this study may improve postoperative care, support earlier clinical intervention, reduce complications, and help healthcare teams provide safer recovery pathways for surgical patients.

DETAILED DESCRIPTION:
Hospital readmissions are well established as key indicators of healthcare quality, particularly in the postoperative setting. Unplanned readmissions often reflect complications that were not fully predicted or adequately managed, generating substantial financial and clinical burden for health systems. In the United States, 3.8 million adult readmissions occurred within 30 days in 2018, with an average cost of US$15,200 per event. In Brazil, similarly high readmission rates have been reported, with 13.4% of more than 22,000 hospitalizations resulting in return visits, largely due to hospital infection, obstructive sleep apnea, and cardiac arrhythmias. Sleep disturbances-including obstructive sleep apnea-are among the most significant contributors to postoperative complications and readmissions. They delay recovery, increase pain sensitivity, impair cognition, and elevate cardiovascular risk. Vascular comorbidities such as hypertension, diabetes, and hyperlipidemia further worsen outcomes by increasing the likelihood of ischemic events, impaired wound healing, and respiratory instability. Understanding how physiologic, behavioral, and sleep-related variables interact to influence postoperative recovery is essential for designing early detection and prevention strategies.

Artificial intelligence (AI) has shown increasing promise in predicting clinical deterioration and identifying high-risk patients across multiple surgical fields. A recent systematic review of 26 studies demonstrated that AI-based models-including natural language processing, classical machine-learning algorithms, and deep learning methods-can accurately predict hospital readmissions following major surgery. However, most available datasets do not combine preoperative, intraoperative, postoperative, and continuous physiologic signals collected in real time from wearable devices, representing a major gap in the literature. This prospective cohort study aims to address this gap by integrating high-resolution physiologic and behavioral data captured from wearable devices-specifically smartwatches and smart rings-into a unified perioperative database, with the overarching goal of developing AI models capable of predicting unplanned hospital readmissions within 30 days after surgery.

The study seeks to build a comprehensive database of patients undergoing medium- to large-scale elective surgeries, capturing physiologic and behavioral data from wearables and multiparametric monitors during the pre- and post-operative periods, including continuous monitoring in the first 48 hours of intensive care when indicated. Data collection will include continuous wearable monitoring via a web-based interface developed by CETELI/UFAM, pre- and post-operative clinical assessments, laboratory tests, imaging studies, pulmonary function evaluations, polysomnography, and validated sleep questionnaires. The study will evaluate correlations between physiologic and sleep-related variables derived from smartwatches and smart rings and the risk of hospital readmission.

Additionally, the study will develop applications for smartwatch and smart ring use in perioperative data capture and employ machine learning approaches-including deep architectures such as causal convolutional networks and recurrent neural networks, as well as classical methods such as support vector machines and decision trees-to predict hospital readmissions. Associations between wearable-derived sleep parameters and 30-day readmission risk will be analyzed, pre- and post-operative sleep data will be correlated with polysomnography and questionnaire results, and sleep quality will be compared between preoperative and post-operative periods.

This research is conducted through a multidisciplinary collaboration between the Hospital Universitário Getúlio Vargas (HUGV-UFAM/Ebserh), and the Center for Research and Development in Electronic and Information Technology (CETELI/UFAM). CETELI will be responsible for developing the data-collection software, storage architecture, and predictive algorithms, while clinical oversight, recruitment, and protocol execution will be led by HUGV.

Beyond scientific relevance, this project has significant practical importance. In geographically complex regions such as the Amazon, continuous remote monitoring using wearable devices can enhance follow-up, reduce disparities in access to postoperative care, and enable earlier identification of complications. Integrating AI-based prediction models with hospital workflows may ultimately reduce costs, optimize patient flow, and improve the safety and quality of surgical care.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age;
* Hospitalization for medium and/or large elective surgery at HUGV;
* Conscious and oriented patients who have sufficient understanding to answer questionnaires and use wearable devices for the study;
* Have minimal skills in the use of wearable technologies;
* Patients who have agreed to participate voluntarily in the research by signing the Informed Consent Form (ICF).

Non-inclusion Criteria:

* Presence of tattoos or any other skin condition (skin pathologies or skin diseases such as vitiligo, lupus, and atopic dermatitis, among others) that affects the area of the wrist or finger where the wearable sensors are located;
* Presence of any type of sensitivity or allergic reaction, of any degree, to the materials of the wearables (smartwatch and smartring);
* Pregnant and lactating women;
* Participants with implantable cardiac devices, such as pacemakers, cardioverter defibrillators, and resynchronization devices;
* Participants in drugs abuse;

Exclusion Criteria:

* Severe medical conditions and decompensations prior to surgery;
* Patients who die before hospital discharge;
* Patients with an expected postoperative hospital stay of more than 10 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients scheduled for medium- and large-scale elective surgeries at the Hospital Universitário Getúlio Vargas, a tertiary referral center in Amazonas. Patients are initially evaluated at the affiliated outpatient clinic, Ambulatório Araújo Lima. Eligible individuals will be invited to participate during preoperative consultations with the attending surgeon, approximately 15 days before hospital admission. Study procedures, information delivery, and informed consent will be conducted by the surgical specialists responsible for outpatient care.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
30-day hospital readmission | Within 30 days post-surgery
  Occurrence of any unplanned hospital readmission within 30 days after discharge following medium- and large-scale surgical procedures. The outcome is binary (Yes/No).

SECONDARY OUTCOMES:
Length of hospital stay | From hospital admission through hospital discharge, up to postoperative day 10
  Total number of days from hospital admission to discharge following the surgical procedure.
Need for reoperation | Up to 30 days after surgery
  Any surgical reintervention required during hospitalization or within the 30-day post-operative period.
Number of Participants With Surgical Site Infection | Up to 30 days post-surgery (or up to hospital discharge if earlier)
30-day mortality | Up to 30 days post-surgery
  All-cause death occurring within 30 days after the surgical procedure.
Subjective Sleep Quality Assessed by the Pittsburgh Sleep Quality Index (PSQI) Total Score | Pre-operative baseline (2 days before admission) and post-operative follow-up at approximately 21-22 days after surgery (±3 days).
  Subjective sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI) total score, which ranges from 0 to 21, with higher scores indicating worse sleep quality.
Insomnia Severity Assessed by the Insomnia Severity Index (ISI) Total Score | Pre-operative baseline (2 days before hospital admission) and post-operative follow-up at approximately 21-22 days after surgery
  Insomnia severity will be assessed using the Insomnia Severity Index (ISI) total score, which ranges from 0 to 28, with higher scores indicating more severe insomnia
Risk of Sleep-Disordered Breathing Assessed by the Neck, Obesity, Snoring, Age, Sex (NoSAS) Score | Pre-operative baseline (2 days before hospital admission) and post-operative follow-up at approximately 21-22 days after surgery
  Risk of sleep-disordered breathing will be assessed using the Neck, Obesity, Snoring, Age, Sex (NoSAS) score, which ranges from 0 to 17, with higher scores indicating a higher risk of sleep-disordered breathing.
Daytime Sleepiness Assessed by the Epworth Sleepiness Scale (ESS) Total Score | Pre-operative baseline (2 days before hospital admission) and post-operative follow-up at approximately 21-22 days after surgery (±3 days)
  Daytime sleepiness will be assessed using the Epworth Sleepiness Scale (ESS) total score, which ranges from 0 to 24, with higher scores indicating greater daytime sleepiness.
Total Sleep Time Assessed by Polysomnography | Pre-operative baseline (2 days before hospital admission) and post-operative follow-up at approximately 21-22 days after surgery
  Total sleep time measured in minutes using overnight polysomnography.
Sleep Efficiency Assessed by Polysomnography | Pre-operative baseline (2 days before hospital admission) and post-operative follow-up at approximately 21-22 days after surgery
  Sleep efficiency measured as a percentage (%) using overnight polysomnography.
Sleep Latency Assessed by Polysomnography | Pre-operative baseline (2 days before hospital admission) and post-operative follow-up at approximately 21-22 days after surgery
  Sleep latency measured in minutes using overnight polysomnography.
Wake After Sleep Onset Assessed by Polysomnography | Pre-operative baseline (2 days before hospital admission) and post-operative follow-up at approximately 21-22 days after surgery
  Wake after sleep onset measured in minutes using overnight polysomnography.
Apnea-Hypopnea Index Assessed by Polysomnography | Pre-operative baseline (2 days before hospital admission) and post-operative follow-up at approximately 21-22 days after surgery
  Apnea-Hypopnea Index (AHI), measured as the number of events per hour of sleep using overnight polysomnography. Higher values indicate more severe sleep-disordered breathing

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elizete de Almeida Araújo, Doctor of Health Science, Study Director — Getúlio Vargas University Hospital; Marly Guimarães Fernandes Costa, Study Director — Federal University of Amazonas; Robson Luís Oliveira de Amorim, Principal Investigator — Getúlio Vargas University Hospital; Caio Eduardo Rodrigues Falcão, Study Chair — Getúlio Vargas University Hospital; Cícero Ferreira Fernandes Costa Filho, Study Chair — Federal University of Amazonas; José Corrêa Lima Netto, Study Chair — Getúlio Vargas University Hospital
Locations (1):
- Getúlio Vargas University Hospital, Manaus, Amazonas, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iucif N Jr, Rocha JS. [Study of inequalities in hospital mortality using the Charlson comorbidity index]. Rev Saude Publica. 2004 Dec;38(6):780-6. doi: 10.1590/s0034-89102004000600005. Epub 2004 Dec 10. Portuguese. PMID 15608895
- [Background] Duarte RL, Magalhaes-da-Silveira FJ, Oliveira-E-Sa TS, Silva JA, Mello FC, Gozal D. Obstructive Sleep Apnea Screening with a 4-Item Instrument, Named GOAL Questionnaire: Development, Validation and Comparative Study with No-Apnea, STOP-Bang, and NoSAS. Nat Sci Sleep. 2020 Jan 23;12:57-67. doi: 10.2147/NSS.S238255. eCollection 2020. PMID 32158294
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Pedro VD, Menna Barreto SS, Johns MW. Portuguese-language version of the Epworth sleepiness scale: validation for use in Brazil. J Bras Pneumol. 2009 Sep;35(9):877-83. doi: 10.1590/s1806-37132009000900009. English, Portuguese. PMID 19820814
- [Background] Yanagimori M, Fernandes MD, Grad GF, Monare AB, Garcia BMSP, Rosanelli I, Mariano PMMS, Drummond SPA, O'Driscoll DM, Edwards BA, Lorenzi-Filho G, Genta PR. Abbreviated versions of the insomnia severity index to screen for comorbid insomnia among obstructive sleep apnea patients. Sleep Med. 2025 Feb;126:19-24. doi: 10.1016/j.sleep.2024.11.035. Epub 2024 Nov 26. PMID 39615273
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Dartora EG, Miozzo IC, de Barba ME, Barreto SS. Validation of the Brazilian Portuguese version of the Pittsburgh Sleep Quality Index. Sleep Med. 2011 Jan;12(1):70-5. doi: 10.1016/j.sleep.2010.04.020. Epub 2010 Dec 9. PMID 21145786
- [Background] Hegab Z, Gibbons S, Neyses L, Mamas MA. Role of advanced glycation end products in cardiovascular disease. World J Cardiol. 2012 Apr 26;4(4):90-102. doi: 10.4330/wjc.v4.i4.90. PMID 22558488
- [Background] Vistoli G, De Maddis D, Cipak A, Zarkovic N, Carini M, Aldini G. Advanced glycoxidation and lipoxidation end products (AGEs and ALEs): an overview of their mechanisms of formation. Free Radic Res. 2013 Aug;47 Suppl 1:3-27. doi: 10.3109/10715762.2013.815348. PMID 23767955
- [Background] Atzeni IM, van de Zande SC, Westra J, Zwerver J, Smit AJ, Mulder DJ. The AGE Reader: A non-invasive method to assess long-term tissue damage. Methods. 2022 Jul;203:533-541. doi: 10.1016/j.ymeth.2021.02.016. Epub 2021 Feb 23. PMID 33636313
- [Background] Amorim RL, Oliveira LM, Malbouisson LM, Nagumo MM, Simoes M, Miranda L, Bor-Seng-Shu E, Beer-Furlan A, De Andrade AF, Rubiano AM, Teixeira MJ, Kolias AG, Paiva WS. Prediction of Early TBI Mortality Using a Machine Learning Approach in a LMIC Population. Front Neurol. 2020 Jan 24;10:1366. doi: 10.3389/fneur.2019.01366. eCollection 2019. PMID 32038454
- [Background] Hale AT, Stonko DP, Lim J, Guillamondegui OD, Shannon CN, Patel MB. Using an artificial neural network to predict traumatic brain injury. J Neurosurg Pediatr. 2019 Feb 1;23(2):219-226. doi: 10.3171/2018.8.PEDS18370. Epub 2018 Nov 2. PMID 30485240
- [Background] Fares MY, Liu HH, da Silva Etges APB, Zhang B, Warner JJP, Olson JJ, Fedorka CJ, Khan AZ, Best MJ, Kirsch JM, Simon JE, Sanders B, Costouros JG, Zhang X, Jones P, Haas DA, Abboud JA; Avant-Garde Health and Codman Society Value-Based Care Group. Utility of Machine Learning, Natural Language Processing, and Artificial Intelligence in Predicting Hospital Readmissions After Orthopaedic Surgery: A Systematic Review and Meta-Analysis. JBJS Rev. 2024 Aug 22;12(8). doi: 10.2106/JBJS.RVW.24.00075. eCollection 2024 Aug 1. PMID 39172864
- [Background] Shameer K, Johnson KW, Yahi A, Miotto R, Li LI, Ricks D, Jebakaran J, Kovatch P, Sengupta PP, Gelijns S, Moskovitz A, Darrow B, David DL, Kasarskis A, Tatonetti NP, Pinney S, Dudley JT. PREDICTIVE MODELING OF HOSPITAL READMISSION RATES USING ELECTRONIC MEDICAL RECORD-WIDE MACHINE LEARNING: A CASE-STUDY USING MOUNT SINAI HEART FAILURE COHORT. Pac Symp Biocomput. 2017;22:276-287. doi: 10.1142/9789813207813_0027. PMID 27896982
- [Background] Min X, Yu B, Wang F. Predictive Modeling of the Hospital Readmission Risk from Patients' Claims Data Using Machine Learning: A Case Study on COPD. Sci Rep. 2019 Feb 20;9(1):2362. doi: 10.1038/s41598-019-39071-y. PMID 30787351
- [Background] Majumder S, Mondal T, Deen MJ. Wearable Sensors for Remote Health Monitoring. Sensors (Basel). 2017 Jan 12;17(1):130. doi: 10.3390/s17010130. PMID 28085085
- [Background] Rumalla K, Srinivasan VM, Gaddis M, Kan P, Lawton MT, Burkhardt JK. Readmission following extracranial-intracranial bypass surgery in the United States: nationwide rates, causes, risk factors, and volume-driven outcomes. J Neurosurg. 2020 Nov 6;135(2):431-439. doi: 10.3171/2020.6.JNS202117. Print 2021 Aug 1. PMID 33157529
- [Background] Li Z, Armstrong EJ, Parker JP, Danielsen B, Romano PS. Hospital variation in readmission after coronary artery bypass surgery in California. Circ Cardiovasc Qual Outcomes. 2012 Sep 1;5(5):729-37. doi: 10.1161/CIRCOUTCOMES.112.966945. Epub 2012 Sep 4. PMID 22949489
- [Background] Silva RAGE, Borgomoni GB, de Freitas FL, Maia ADS, Farias do Vale Junior C, Pereira EDS, Silvestre LGI, Dallan LRP, Lisboa LA, Dallan LAO, Jatene FB, Mejia OAV; grupo de estudos REPLICCAR. Predictors of 30-Day Hospital Readmission Following CABG in a Multicenter Database: A Cross-Sectional Study. Arq Bras Cardiol. 2024 Sep 6;121(9):e20230768. doi: 10.36660/abc.20230768. eCollection 2024. English, Portuguese. PMID 39258643
- [Background] Scalzitti NJ, O'Connor PD, Nielsen SW, Aden JK, Brock MS, Taylor DM, Mysliwiec V, Dion GR. Obstructive Sleep Apnea is an Independent Risk Factor for Hospital Readmission. J Clin Sleep Med. 2018 May 15;14(5):753-758. doi: 10.5664/jcsm.7098. PMID 29734972
- [Background] Lan T, Liao YH, Zhang J, Yang ZP, Xu GS, Zhu L, Fan DM. Mortality and Readmission Rates After Heart Failure: A Systematic Review and Meta-Analysis. Ther Clin Risk Manag. 2021 Dec 7;17:1307-1320. doi: 10.2147/TCRM.S340587. eCollection 2021. PMID 34908840
- [Background] Psotka MA, Fonarow GC, Allen LA, Joynt Maddox KE, Fiuzat M, Heidenreich P, Hernandez AF, Konstam MA, Yancy CW, O'Connor CM. The Hospital Readmissions Reduction Program: Nationwide Perspectives and Recommendations: A JACC: Heart Failure Position Paper. JACC Heart Fail. 2020 Jan;8(1):1-11. doi: 10.1016/j.jchf.2019.07.012. Epub 2019 Oct 9. PMID 31606360
- [Background] Jencks SF, Williams MV, Coleman EA. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Apr 2;360(14):1418-28. doi: 10.1056/NEJMsa0803563. PMID 19339721